CLINICAL TRIAL: NCT04058548
Title: Clinical Utility of the 1-minute Sit to Stand Test as a Measure of Submaximal Exercise Tolerance in Patients With Cystic Fibrosis During Acute Pulmonary Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jenna Gondelman, Physical Therapist 2, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-P00031139
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; walk test
MeSH Terms: conditions — Cystic Fibrosis | interventions — Walk Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6MWT and STS (Experimental): All participates will receive 6MWT and STS test
  Interventions: Diagnostic Test: Sit to stand test

INTERVENTIONS:
Diagnostic Test: Sit to stand test — Participants will complete a sit to stand test in addition to a 6 minute walk test
  Other Names: 6 minute walk test

SUMMARY:
The aim of this study is to assess whether the 1 minute Sit to Stand (STS) test can be used as a measure of submaximal endurance during a pulmonary exacerbation of Cystic Fibrosis (CF) for patients in the acute care setting. We hypothesize that if the STS test is a valid measure of submaximal cardiovascular endurance, it will moderately correlate with 6 minute walk distance (6MWD).

ELIGIBILITY:
Inclusion Criteria:

* patients age 6-35 with cystic fibrosis who are admitted for a pulmonary exacerbation and receive ongoing physical therapy throughout their admission.

Exclusion Criteria:

* patients with cystic fibrosis who are under the age of 6,
* patients with cystic fibrosis who are not admitted for a pulmonary exacerbation,
* patients with cystic fibrosis who are not being followed regularly by physical therapy (>5x/week) throughout their inpatient admission,
* patients with cystic fibrosis who are unable to follow instructions for standardized testing,
* patients with cystic fibrosis who are not medically stable to participate in submaximal exercise testing.
* patients whose inpatient admission is anticipated to be <1 week.
* Patients who are readmitted to the hospital within the year will not be included in the study more than once.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
1-minute STS repetitions: | 1 minute
  Number of STS completed
1 minute STS power: | 1 minute
  number of STS completed in 1 minute multiplied by bodyweight in pounds
6 Minute Walk Distance (6MWD): | 6 minutes
  total distance in feet completed during test
6MWT power | 6 minutes
  total distance in feet multiplied by bodyweight in pounds

SECONDARY OUTCOMES:
Heart rate | 1 minute
  beats per minute
Oxygen saturation | 1-6 minutes
  percentage via pulse oximetry
Respiratory rate | 1-6 min
  breaths per minute
Rating of perceived exertion | 6 minutes
  rating via Borg scale for perceived exertion: 0-10 with 0 being no breathlessness and 10 being maximal breathlessness

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Gondelman, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrade Lima C, Dornelas de Andrade A, Campos SL, Brandao DC, Mourato IP, Britto MCA. Six-minute walk test as a determinant of the functional capacity of children and adolescents with cystic fibrosis: A systematic review. Respir Med. 2018 Apr;137:83-88. doi: 10.1016/j.rmed.2018.02.016. Epub 2018 Feb 26. PMID 29605218
- [Background] Gruet M, Peyre-Tartaruga LA, Mely L, Vallier JM. The 1-Minute Sit-to-Stand Test in Adults With Cystic Fibrosis: Correlations With Cardiopulmonary Exercise Test, 6-Minute Walk Test, and Quadriceps Strength. Respir Care. 2016 Dec;61(12):1620-1628. doi: 10.4187/respcare.04821. Epub 2016 Nov 15. PMID 27899540
- [Background] Radtke T, Puhan MA, Hebestreit H, Kriemler S. The 1-min sit-to-stand test--A simple functional capacity test in cystic fibrosis? J Cyst Fibros. 2016 Mar;15(2):223-6. doi: 10.1016/j.jcf.2015.08.006. Epub 2015 Sep 9. PMID 26363563
- [Background] Okuro RT, de Oliveira Ribeiro MA, Ribeiro JD, Minsky RC, Schivinski CI. Alternative Indexes to Estimate the Functional Capacity From the 6-Minute Walk Test in Children and Adolescents With Cystic Fibrosis. Respir Care. 2017 Mar;62(3):324-332. doi: 10.4187/respcare.04625. Epub 2017 Jan 3. PMID 28049743
- [Background] Vaidya T, de Bisschop C, Beaumont M, Ouksel H, Jean V, Dessables F, Chambellan A. Is the 1-minute sit-to-stand test a good tool for the evaluation of the impact of pulmonary rehabilitation? Determination of the minimal important difference in COPD. Int J Chron Obstruct Pulmon Dis. 2016 Oct 19;11:2609-2616. doi: 10.2147/COPD.S115439. eCollection 2016. PMID 27799759